CLINICAL TRIAL: NCT04784676
Title: Internal Fit Evaluation of Indirect Restorations Fabricated From CAD/CAM Composite Blocks Versus Ceramic Blocks in Badly Broken Teeth Using Cone Beam CT (CBCT)
Brief Title: Internal Fit Evaluation of Indirect Restorations Using Cone Beam CT (CBCT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study is ended
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shereen Hafez Ibrahim Mohamed, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8-3-19
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Indirect Restoration of Badly Broken Vital Teeth
Keywords: randomized clinical trial; internal adaptation; CAD/CAM composite restoration; all ceramic restoration; E-max CAD; CAD/CAM milling system; CAD/CAD; composite; inlays; onlays; cone beam CT; CBCT

STUDY DESIGN:
Intervention Model Description: randomized clinical trial parallel group, two arms, superiority trial, allocation ratio 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: allocation concealment by opaque sealed envelopes, the participants and assessors were blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nanohybrid composite blocks (Experimental): nanohybrid composite CAD/CAM blocks
  Interventions: Other: restoration
- ceramic blocks (Active Comparator): ceramic CAD/CAM blocks emax
  Interventions: Other: restoration

INTERVENTIONS:
Other: restoration — indirect restoration

SUMMARY:
this study was conducted to evaluate the internal fit of indirect restoration fabricated from CAD/CAM composite blocks versus ceramic blocks in badly broken vital teeth using cone beam CT

DETAILED DESCRIPTION:
two parallel groups (n=42 restorations), patient having badly broken vital teeth minimum of two remaining wall will be randomly enrolled in this trial and receive restoration fabricated either from Grandio composite blocks or E-max ceramic blocks. internal fit evaluation of the fabricated restoration over their corresponding casts will be performed using cone beam CT just prior cementation of the restorations. data will be collected and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients with badly broken vital teeth young adult males or females (20-50 years) good oral hygeine cooperative patients approving to participate in the study

Exclusion Criteria:

* patients with acompromised medical history severe or active periodontal disease severe medical complications lack of compliance

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
internal fit evaluation | on cast before delivery
  in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Shereen H Ibrahim, PhD, Principal Investigator — associate professor of conservative Dentistry, faculty of dentistry Cairo university Egypt
Locations (1):
- faculty of dentistry, Cairo University, Cairo, Please Select..., Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim SH, Amr H, Hassan AA, Elzohairy A. Internal fit evaluation of indirect restorations fabricated from CAD/CAM composite blocks versus ceramic blocks in badly broken teeth using cone beam CT (CBCT): double-blinded randomized clinical trial. Heliyon. 2022 May 19;8(5):e09466. doi: 10.1016/j.heliyon.2022.e09466. eCollection 2022 May. PMID 35647344